CLINICAL TRIAL: NCT03501160
Title: Socially Inappropriate Behaviour in People With First Episode Psychosis: A Caregivers' Perspective
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chan Cheuk Yin, Registered Nurse (Psychiatric), Hospital Authority, Hong Kong
Other Study IDs: Joint CUHK-NTEC CREC 2018.079
Record Dates: First submitted 2018-04-01; First posted 2018-04-18 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: First Episode Psychosis
Keywords: Regressive behaviors; Childish behaviors; Socially Inappropriate Behaviors; Qualitative study; Schizophrenic spectrum disorder; First episode psychosis; Caregiving experience; Caregiving distress

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Face-to face semi-structured in-depth interview — Face-to face semi-structured in-depth interview will be arranged in order to explore the inappropriate social behavior and caregiver stress from caregivers. The interview will be guided by a semi-structured interview guide which specially designed for exploring clinical picture of inappropriate social and affectionate behavior and caregiving distress. The interview guide mainly consisted of specific questions and open-ended questions that encourage the subjects to talk freely in relevant topics during interview. Demographic data was also collected in the beginning of interview. Each interview will be conducted around 60 minutes until data saturated. The interview will be audio-taped with informed consent from subjects.

SUMMARY:
Social impairment is one of the core symptoms in first episode psychosis (FEP). Despite negative symptoms and social cognition impairment found in patient suffering from FEP, clinicians occasionally identified socially inappropriate behaviours (SIB) after onset and stabilization of psychotic disorder. It is also uncommon that some caregivers often complain about their relatives with psychosis of embarrassing and immature behaviour. SIB mainly observed in form of excessive emotional expression, childish behaviour and regressive behaviour. There is limited research focusing on this inadequate behavioural pattern in patient with first episode psychosis recently. It was worth investigating this phenomenon and gain more understanding in other comorbidity symptoms and caregiving distress arisen from this. Psychometric tests and validated assessment tools are well-developed for measuring positive symptoms, negative symptoms, neurocognitive deficits and social cognition impairment in schizophrenic patients but none of them is useful specifically for assessing SIB, and not to mention, from carer's perspective. It could be an obstacle for clinicians to investigate the phenomena of the prevalence and the impact on family in real life without any validated assessment tools or questionnaires. This qualitative study aims to identify the SIB in patients with FEP and to explore the caregiving experience and distress. Hopefully, this study may help designing a questionnaire for future exploration on this topic.

DETAILED DESCRIPTION:
Study Design

This study will be conducted in descriptive qualitative design. Descriptive qualitative design is an eclectic and pragmatic approach. It presents comprehensive summaries of a phenomenon or events in everyday language. It studies a phenomenon to discover patterns and themes about life events intensely. Meanings of the data provided by informants should be kept as much as possible in any interpretation of the researcher. It helps to in-depth understand the experiences of caring individuals with first episode psychosis in Hong Kong. It also allows them to express their observed socially inappropriate behaviors and perceived burdens and coping strategies in their own words. It allows researches to focus on discovering the experiences and gaining insights from informants regarding a poorly understood phenomenon and develop questionnaires or interventions.

Sampling

Purposive sampling will be employed in this study. Purposive sampling allows rich and in-depth data collection as researcher purposely selecting subjects who are judged to be suitable in the population or particularly knowledgeable about the issues under study. It is particular well suited to this study as it provides a systematic way of exploring the full picture of the observed phenomenon. Using homogeneous purposive sampling can ensure selecting samples for having a shared characteristic or set of characteristics and focusing on one specific subgroup in which all the sample members are similar in a particular level or hierarchy.

The subjects will be recruited from Alice Ho Miu Ling Nethersole Hospital (AHNH) and North District Hospital (NDH) psychiatric specialist out-patient clinic. The psychiatrists working in Early Assessment Services for Young People with psychosis (EASY) team will refer the suitable Chinese cases after granted the agreement from potential subjects. The Inclusion criteria framed all target subjects were Hong Kong primary caregivers whose offspring was primary diagnosed of schizophrenic spectrum disorder with social inappropriate behavior after onset of illness. The patient should be under active care by EASY team. The cases of bipolar affective disorder and drug induced psychosis should be excluded from the study. In addition, the cases of active substance abuse and presenting active psychotic symptoms were also not suitable for the study.

Study Population Description

Socially inappropriate behavior was occasionally identified by clinicians in patient with first episode psychosis. SIB was mainly observed as social inappropriate affectionate behavior, childish behavior and regressive behavior. Clinicians observed some patient became excessively dependent on family members and displayed intimate physical contact towards family members. Such socially inappropriate behaviors may explain by frontal lobe dysfunction or deficits in theory of mind.

Socially inappropriate behaviour, as well as social disinhibition, is defined as inappropriate behaviours in term of verbal, physical or sexual acts which reflect a loss of inhibition or an inability to conform to social or cultural behavioural norms. The broad definition of SIB is regarded as physical actions with intimate or sexual behaviours which acting impulsively in motor and verbal expression. Also, SIB is also descried as a behavioural syndrome characterized by immaturity and insensitivity towards others. Research study showed SIB could be assumed to result from deficits in theory of mind as patient failed to understanding of other's mind and perspective. Various psychiatric and neurologic disorders are notable for further developing of socially inappropriate behaviours. Frontal lobe dysfunction, frontal lobe lesions, traumatic brain injury, Tourette's syndrome and frontotemporal dementia were found correlated to the development of socially inappropriate behaviours. The affected patients are unable to correctly identify moral transgressions or having impairment in judgement in their actual behaviours, excessive emotionally based acts and sexual misbehaviours.

Research studies indicated evidence in frontal lobe dysfunction is one of the major causes of SIB in the pathogenesis of schizophrenic spectrum disorder. The schizophrenic patient who suffered from frontal lobe damage demonstrated dramatic personality change, cognitive impairment and negative symptoms. The frontal system damage induced specific impairment of deficits in various aspects especially causing impulsive acts, inappropriate activities, excessive emotional expressions and childish behaviours. It is commonly to find patient shown declining in cognitive functioning, social impairment, poor motivation, lack of responsibility and impaired judgement in related to frontal lobe dysfunction.

Data Collection

Face-to face semi-structured in-depth interview will be arranged in order to explore the inappropriate social behavior and caregiver stress from caregivers. The interview will be guided by a semi-structured interview guide which specially designed for exploring clinical picture of inappropriate social and affectionate behavior and caregiving distress. The interview guide mainly consisted of specific questions and open-ended questions that encourage the subjects to talk freely in relevant topics during interview. Demographic data was also collected in the beginning of interview. Each interview will be conducted around 60 minutes until data saturated. The interview will be audio-taped with informed consent from subjects. The interview will be audio-taped and being transcribed into verbatim in text material for data analysis.

Data analysis

Data collected in the interview was audio taped and being transcribed into verbatim in text material for data analysis. Content analysis is used for analyzing the content of the collected data. It is used for analyzing the numerous findings to identify prominent themes and patterns among all collected data. It is commonly known as breaking down collected data into smaller units and grouping the similar content and concept into a sub-group with specific coding and naming. Phases and key words identified in the content of collected data which shared the common ground and meaning were interpreted and divided into related themes in order to disseminate the findings in category scheme. It determines the trends and relationship of reality by systematic coding and categorizing approach. Verbatim and related narrative materials were reviewed repeatedly by principal investigator in order to identify the underlying themes accurately and precisely.

Ethical Consideration

The study was governed and monitored by NTEC-CUHK Joint CREC. Potential subjects were invited purposively to attend the interview with full disclosure of the study. Written informed consent must be obtained from the subjects before the interview. The consent form clearly stated the essential information of study and the rights of being a research subject in Chinese. Subjects had freedom to refuse joining the study and answering questions from researchers. Subjects had the right to withdraw from the study at any time. All data and information collected was regarded as confidential and strictly accessible by responding researchers only. All data collected will be encrypted with password (electronic documents) and placed in safety place with double lock (written documents). All data and information collected in the study including audio-tape recordings and the verbatim materials will be destroyed after the completion of the study. This study do not involve any treatment or procedure differ from current treatment practice to subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Active Chinese case in psychiatric specialist out-patient clinic
2. Suffering from schizophrenic spectrum disorder (ICD-10)
3. Showing socially inappropriate behavior after onset and stabilization of schizophrenic spectrum disorder

Exclusion Criteria:

1. Case of bipolar affective disorder, drug induced psychosis and intellectual disability
2. Case of active substance abuse
3. Case of presenting active psychotic symptoms

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Social impairment is one of the core symptoms in first episode psychosis and a part of its diagnostic criteria. Social impairment not only affects families and working performance but also creates distress and disharmony in social interactions and relationships. Despite of negative symptoms and social cognitive impairment found in patient suffering from first episode psychosis, clinicians occasionally identified socially inappropriate affectionate behavior after onset of psychotic disorder. Socially inappropriate behavior was mainly observed as social inappropriate affectionate behavior, childish behavior and regressive behavior. Clinicians observed some patient became excessively dependent on family members and displayed intimate physical contact towards family members.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Socially inappropriate behavior in patients with first episode psychosis and its related prevailing caregiving stress and burdens. | 12 Months
  To identify and assess the clinical pictures of socially inappropriate behavior in first episode psychosis and its impact and related caregiving stress from caregivers' perspective by using face-to face semi-structured in-depth interview.
  This piece of study would explore the socially inappropriate behavior in patients with first episode psychosis. This study was expected to provide a descriptive summary and further understanding on the phenomenon interested. It would hope to arouse social attention and provide insight in future planning of social and healthcare resources in community regarding the prevailing burdens and caregiving stress perceived by caregivers of individuals who diagnosed first episode psychosis with socially inappropriate behavior in Hong Kong.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - North District Hospital, Hospital Authority, Sheung Shui
  - Alice Ho Miu Ling Nethersole Hospital, Hospital Authority, HKSAR, Tai Po

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arciniegas DB, Wortzel HS. Emotional and behavioral dyscontrol after traumatic brain injury. Psychiatr Clin North Am. 2014 Mar;37(1):31-53. doi: 10.1016/j.psc.2013.12.001. PMID 24529422
- [Background] Bratlien U, Oie M, Lien L, Agartz I, Lie Romm K, Vaskinn A, Ueland T, Andreassen OA, Melle I. Social dysfunction in first-episode psychosis and relations to neurocognition, duration of untreated psychosis and clinical symptoms. Psychiatry Res. 2013 May 15;207(1-2):33-9. doi: 10.1016/j.psychres.2012.10.010. Epub 2012 Nov 13. PMID 23153893
- [Background] Breitborde NJ, Kleinlein P, Srihari VH. Self-determination and first-episode psychosis: associations with symptomatology, social and vocational functioning, and quality of life. Schizophr Res. 2012 May;137(1-3):132-6. doi: 10.1016/j.schres.2012.02.026. Epub 2012 Mar 22. PMID 22445463
- [Background] Breitborde NJ, Srihari VH, Woods SW. Review of the operational definition for first-episode psychosis. Early Interv Psychiatry. 2009 Nov;3(4):259-65. doi: 10.1111/j.1751-7893.2009.00148.x. PMID 22642728
- [Background] Chang WC, Lau CFC, Chan SSI, Hui CLM, Chan SKW, Lee EHM, Lin J, Chen EYH. Premorbid, clinical and cognitive correlates of primary negative symptoms in first-episode psychosis. Psychiatry Res. 2016 Aug 30;242:144-149. doi: 10.1016/j.psychres.2016.05.045. Epub 2016 Jun 1. PMID 27280524
- [Background] Chen ES, Chang WC, Hui CL, Chan SK, Lee EH, Chen EY. Self-stigma and affiliate stigma in first-episode psychosis patients and their caregivers. Soc Psychiatry Psychiatr Epidemiol. 2016 Sep;51(9):1225-31. doi: 10.1007/s00127-016-1221-8. Epub 2016 Apr 27. PMID 27118543
- [Background] Compton, M. T., & Broussard, B. (2009). The first episode of psychosis: A guide for patients and their families. Oxford: Oxford University Press
- [Background] Cornblatt BA, Carrion RE, Addington J, Seidman L, Walker EF, Cannon TD, Cadenhead KS, McGlashan TH, Perkins DO, Tsuang MT, Woods SW, Heinssen R, Lencz T. Risk factors for psychosis: impaired social and role functioning. Schizophr Bull. 2012 Nov;38(6):1247-57. doi: 10.1093/schbul/sbr136. Epub 2011 Nov 10. PMID 22080497
- [Background] Corrigan, P. W., & Watson, A. C. (2002). The paradox of self-stigma and mental illness. Clinical Psychology: Science & Practice, 9, 35-53.
- [Background] Cowen, P., Harrison, P., & Burns, T. (2012). Shorter Oxford textbook of psychiatry. Oxford: Oxford University Press.
- [Background] Cressman VL, Schobel SA, Steinfeld S, Ben-David S, Thompson JL, Small SA, Moore H, Corcoran CM. Anhedonia in the psychosis risk syndrome: associations with social impairment and basal orbitofrontal cortical activity. NPJ Schizophr. 2015 Jul 15;1:15020. doi: 10.1038/npjschz.2015.20. eCollection 2015. PMID 27336033
- [Background] Cuesta MJ, Garcia de Jalon E, Campos MS, Ibanez B, Sanchez-Torres AM, Peralta V. Duration of untreated negative and positive symptoms of psychosis and cognitive impairment in first episode psychosis. Schizophr Res. 2012 Nov;141(2-3):222-7. doi: 10.1016/j.schres.2012.08.019. Epub 2012 Sep 16. PMID 22989921
- [Background] Dodell-Feder D, Tully LM, Hooker CI. Social impairment in schizophrenia: new approaches for treating a persistent problem. Curr Opin Psychiatry. 2015 May;28(3):236-42. doi: 10.1097/YCO.0000000000000154. PMID 25768085
- [Background] Eddy CM, Cavanna AE. On being your own worst enemy: an investigation of socially inappropriate symptoms in Tourette syndrome. J Psychiatr Res. 2013 Sep;47(9):1259-63. doi: 10.1016/j.jpsychires.2013.05.019. Epub 2013 Jun 13. PMID 23768869
- [Background] Elo S, Kyngas H. The qualitative content analysis process. J Adv Nurs. 2008 Apr;62(1):107-15. doi: 10.1111/j.1365-2648.2007.04569.x. PMID 18352969
- [Background] Finger EC, Marsh AA, Kamel N, Mitchell DG, Blair JR. Caught in the act: the impact of audience on the neural response to morally and socially inappropriate behavior. Neuroimage. 2006 Oct 15;33(1):414-21. doi: 10.1016/j.neuroimage.2006.06.011. Epub 2006 Aug 7. PMID 16891125
- [Background] Foussias G, Remington G. Negative symptoms in schizophrenia: avolition and Occam's razor. Schizophr Bull. 2010 Mar;36(2):359-69. doi: 10.1093/schbul/sbn094. Epub 2008 Jul 21. PMID 18644851
- [Background] Gee B, Hodgekins J, Fowler D, Marshall M, Everard L, Lester H, Jones PB, Amos T, P Singh S, Sharma V, Freemantle N, Birchwood M. The course of negative symptom in first episode psychosis and the relationship with social recovery. Schizophr Res. 2016 Jul;174(1-3):165-171. doi: 10.1016/j.schres.2016.04.017. Epub 2016 Apr 28. PMID 27131912
- [Background] Gronholm PC, Thornicroft G, Laurens KR, Evans-Lacko S. Mental health-related stigma and pathways to care for people at risk of psychotic disorders or experiencing first-episode psychosis: a systematic review. Psychol Med. 2017 Aug;47(11):1867-1879. doi: 10.1017/S0033291717000344. Epub 2017 Feb 15. PMID 28196549
- [Background] Guastella AJ, Hermens DF, Van Zwieten A, Naismith SL, Lee RS, Cacciotti-Saija C, Scott EM, Hickie IB. Social cognitive performance as a marker of positive psychotic symptoms in young people seeking help for mental health problems. Schizophr Res. 2013 Sep;149(1-3):77-82. doi: 10.1016/j.schres.2013.06.006. Epub 2013 Jul 9. PMID 23845388
- [Background] Ho KK, Lui SS, Hung KS, Wang Y, Li Z, Cheung EF, Chan RC. Theory of mind impairments in patients with first-episode schizophrenia and their unaffected siblings. Schizophr Res. 2015 Aug;166(1-3):1-8. doi: 10.1016/j.schres.2015.05.033. Epub 2015 Jun 3. PMID 26049215
- [Background] Holroyd EE. Chinese cultural influences on parental caregiving obligations toward children with disabilities. Qual Health Res. 2003 Jan;13(1):4-19. doi: 10.1177/1049732302239408. PMID 12564260
- [Background] Hwang, K. K. (1997). Guanxi and mientze: Conflict resolution in Chinese society. Intercultural Communication Studies, 7, 17-42.
- [Background] Jansen JE, Lysaker PH, Harder S, Haahr UH, Lyse HG, Pedersen MB, Trauelsen AM, Simonsen E. Positive and negative caregiver experiences in first-episode psychosis: emotional overinvolvement, wellbeing and metacognition. Psychol Psychother. 2014 Sep;87(3):298-310. doi: 10.1111/papt.12014. Epub 2013 Sep 3. PMID 24038708
- [Background] Jansen JE, Gleeson J, Cotton S. Towards a better understanding of caregiver distress in early psychosis: a systematic review of the psychological factors involved. Clin Psychol Rev. 2015 Feb;35:56-66. doi: 10.1016/j.cpr.2014.12.002. Epub 2014 Dec 12. PMID 25531423
- [Background] Jansen JE, Haahr UH, Harder S, Trauelsen AM, Lyse HG, Buch Pedersen M, Simonsen E. Caregiver distress in first-episode psychosis: the role of subjective appraisal, over-involvement and symptomatology. Soc Psychiatry Psychiatr Epidemiol. 2015 Mar;50(3):371-8. doi: 10.1007/s00127-014-0935-8. Epub 2014 Jul 23. PMID 25053150
- [Background] Kelly G, Brown S, Todd J, Kremer P. Challenging behaviour profiles of people with acquired brain injury living in community settings. Brain Inj. 2008 Jun;22(6):457-70. doi: 10.1080/02699050802060647. PMID 18465387
- [Background] Kidd SA. From social experience to illness experience: reviewing the psychological mechanisms linking psychosis with social context. Can J Psychiatry. 2013 Jan;58(1):52-8. doi: 10.1177/070674371305800110. PMID 23327757
- [Background] Kung, W. W. (2001). Consideration of cultural factors in working with Chinese American families with a mentally ill patient. Families in Society, 82, 97-107.
- [Background] Lau, D. Y. K., & Pang, A. H. T. (2007). Validation of the Chinese version of experience of caregiving inventory in caregivers of persons suffering from severe mental disorders. Hong Kong Journal of Psychiatry, 17(1), 24-32.
- [Background] Lee SJ, Kim KR, Lee SY, An SK. Impaired Social and Role Function in Ultra-High Risk for Psychosis and First-Episode Schizophrenia: Its Relations with Negative Symptoms. Psychiatry Investig. 2017 Mar;14(2):186-192. doi: 10.4306/pi.2017.14.2.186. Epub 2017 Mar 6. PMID 28326117
- [Background] Link, B. G., & Phelan, J. C. (2001). Conceptualizing stigma. Annual Review of Sociology, 27, 363-385.
- [Background] Lokko HN, Stern TA. Regression: Diagnosis, Evaluation, and Management. Prim Care Companion CNS Disord. 2015 May 14;17(3):10.4088/PCC.14f01761. doi: 10.4088/PCC.14f01761. eCollection 2015. No abstract available. PMID 26644947
- [Background] Magilvy JK, Thomas E. A first qualitative project: qualitative descriptive design for novice researchers. J Spec Pediatr Nurs. 2009 Oct;14(4):298-300. doi: 10.1111/j.1744-6155.2009.00212.x. No abstract available. PMID 19796329
- [Background] Mak, W. W. S., & Cheung, R. Y. M. (2008). Affiliate stigma among caregivers of people with mental illness or intellectual disability. Journal of Applied Research in Intellectual Disabilities, 21, 532-545.
- [Background] Mak WW, Cheung RY. Psychological distress and subjective burden of caregivers of people with mental illness: the role of affiliate stigma and face concern. Community Ment Health J. 2012 Jun;48(3):270-4. doi: 10.1007/s10597-011-9422-9. Epub 2011 Jun 17. PMID 21681460
- [Background] Mak WW, Chong ES, Wong CC. Beyond attributions: Understanding public stigma of mental illness with the common sense model. Am J Orthopsychiatry. 2014 Mar;84(2):173-81. doi: 10.1037/h0099373. PMID 24826933
- [Background] McKhann GM, Albert MS, Grossman M, Miller B, Dickson D, Trojanowski JQ; Work Group on Frontotemporal Dementia and Pick's Disease. Clinical and pathological diagnosis of frontotemporal dementia: report of the Work Group on Frontotemporal Dementia and Pick's Disease. Arch Neurol. 2001 Nov;58(11):1803-9. doi: 10.1001/archneur.58.11.1803. PMID 11708987
- [Background] Mercer J. The concept of psychological regression: metaphors, mapping, Queen Square, and Tavistock Square. Hist Psychol. 2011 May;14(2):174-96. doi: 10.1037/a0022710. PMID 21688725
- [Background] Meyer, R. A. & Maccabe, L. R. (2012). Schizophrenia. Medicine, 40(11), 586-590.
- [Background] Millan MJ, Fone K, Steckler T, Horan WP. Negative symptoms of schizophrenia: clinical characteristics, pathophysiological substrates, experimental models and prospects for improved treatment. Eur Neuropsychopharmacol. 2014 May;24(5):645-92. doi: 10.1016/j.euroneuro.2014.03.008. Epub 2014 Apr 4. PMID 24820238
- [Background] Mitsonis C, Voussoura E, Dimopoulos N, Psarra V, Kararizou E, Latzouraki E, Zervas I, Katsanou MN. Factors associated with caregiver psychological distress in chronic schizophrenia. Soc Psychiatry Psychiatr Epidemiol. 2012 Feb;47(2):331-7. doi: 10.1007/s00127-010-0325-9. Epub 2010 Dec 17. PMID 21165597
- [Background] Mo, F. Y., Chung, W. S., Wong, S. W., Chun, D. Y. Y., Wong, K. S., & Chan, S. S. M. (2008). Experience of caregiving in caregivers of patients with first-episode psychosis. East Asian Archives of Psychiatry, 18(3), 101.
- [Background] Ohmuro N, Katsura M, Obara C, Kikuchi T, Sakuma A, Iizuka K, Hamaie Y, Ito F, Matsuoka H, Matsumoto K. Deficits of cognitive theory of mind and its relationship with functioning in individuals with an at-risk mental state and first-episode psychosis. Psychiatry Res. 2016 Sep 30;243:318-25. doi: 10.1016/j.psychres.2016.06.051. Epub 2016 Jul 1. PMID 27434201
- [Background] Osborne-Crowley K, McDonald S. A review of social disinhibition after traumatic brain injury. J Neuropsychol. 2018 Jun;12(2):176-199. doi: 10.1111/jnp.12113. Epub 2016 Sep 30. PMID 27696753
- [Background] Pazvantoğlu, O., Sarısoy, G., Böke, Ö., Aker, A. A., Özturan, D. D., & Ünverdi, E. (2014). The dimensions of caregiver burden in schizophrenia: The role of patients functionality. Düşünen Adam: The Journal of Psychiatry and Neurological Sciences, 27(1), 53-60.
- [Background] Polit, D. F., & Beck, C. T. (2013). Essentials of nursing research: Appraising evidence for nursing practice. Lippincott Williams & Wilkins.
- [Background] Renwick L, Jackson D, Foley S, Owens E, Ramperti N, Behan C, Anwar M, Kinsella A, Turner N, Clarke M, O'Callaghan E. Depression and quality of life in first-episode psychosis. Compr Psychiatry. 2012 Jul;53(5):451-5. doi: 10.1016/j.comppsych.2011.07.003. Epub 2011 Aug 25. PMID 21871616
- [Background] Stuss DT, Gow CA, Hetherington CR. "No longer Gage": frontal lobe dysfunction and emotional changes. J Consult Clin Psychol. 1992 Jun;60(3):349-59. doi: 10.1037//0022-006x.60.3.349. PMID 1619089
- [Background] SUTTELL BJ, PASCAL GR. "Regression" in schizophrenia as determined by performance on the Bender-Gestalt test. J Abnorm Psychol. 1952 Jul;47(3):653-7. doi: 10.1037/h0059987. No abstract available. PMID 12980767
- [Background] Tomlinson E, Onwumere J, Kuipers E. Distress and negative experiences of the caregiving relationship in early psychosis: does social cognition play a role? Early Interv Psychiatry. 2014 Aug;8(3):253-60. doi: 10.1111/eip.12040. Epub 2013 Mar 12. PMID 23489370
- [Background] Vohs JL, Lysaker PH, Francis MM, Hamm J, Buck KD, Olesek K, Outcalt J, Dimaggio G, Leonhardt B, Liffick E, Mehdiyoun N, Breier A. Metacognition, social cognition, and symptoms in patients with first episode and prolonged psychoses. Schizophr Res. 2014 Mar;153(1-3):54-9. doi: 10.1016/j.schres.2014.01.012. Epub 2014 Feb 4. PMID 24503175
- [Background] Walker JL. The use of saturation in qualitative research. Can J Cardiovasc Nurs. 2012 Spring;22(2):37-46. English, French. PMID 22803288
- [Background] Weinberger DR. Schizophrenia and the frontal lobe. Trends Neurosci. 1988 Aug;11(8):367-70. doi: 10.1016/0166-2236(88)90060-4. No abstract available. PMID 2469198
- [Background] Weinberger DR, Berman KF, Zec RF. Physiologic dysfunction of dorsolateral prefrontal cortex in schizophrenia. I. Regional cerebral blood flow evidence. Arch Gen Psychiatry. 1986 Feb;43(2):114-24. doi: 10.1001/archpsyc.1986.01800020020004. PMID 3947207
- [Background] Zhu CY, Lee TM, Li XS, Jing SC, Wang YG, Wang K. Impairments of social cues recognition and social functioning in Chinese people with schizophrenia. Psychiatry Clin Neurosci. 2007 Apr;61(2):149-58. doi: 10.1111/j.1440-1819.2007.01630.x. PMID 17362432